CLINICAL TRIAL: NCT00487955
Title: The Metabolic Contribution of the Human Microbiota to Resting Energy Expenditure
Acronym: A-P-REE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-AH-176-CTIL
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-03

CONDITIONS: Gastritis
Keywords: gastritis; helicobacter pylori; REE; patients with gastritis that refers to helicobacter pylori treatment
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Resting Energy Expenditure examination

SUMMARY:
The purpose of our study is to evaluate the metabolic contribution of the human microbiota to resting energy expenditure

DETAILED DESCRIPTION:
There are now >500 million adult humans in the world who are overweight [body mass index (BMI) of 25.0-29.9 kg/m2] and 250 million who are obese (BMI 30 kg/m2). This growing epidemic threatens both industrialized and developing countries and has been accompanied by worldwide increases in obesity-related disorders, including type II diabetes, hypertension, cardiovascular pathology, and nonalcoholic fatty liver disease. In the United States, 64% of adults are overweight or obese, prompting the Surgeon General to designate this condition as the most important public health challenge of our time.

The worldwide obesity epidemic is stimulating efforts to identify host and environmental factors that affect energy balance. The Human gut contains an immense number of microorganisms, collectively known as the microbiota. This community consists of at least 1013 citizens, is dominated by anaerobic bacteria, and includes 500-1,000 species whose collective genomes are estimated to contain 100 times more genes than our own human genome. The microbiota can be viewed as a metabolic "organ" exquisitely tuned to our physiology that performs functions that we have not had to evolve on our own. These functions include the ability to process otherwise indigestible components of our diet, such as plant polysaccharides, and therefore may have an impact on our energy balance.

Comparisons of the distal gut microbiota of genetically obese mice and their lean littermates, as well as those of obese and lean human volunteers have revealed that obesity is associated with changes in the relative abundance of two dominant bacterial divisions, the Bacteroidetes and the Firmicutes. Turnbaugh et al demonstrated through metagenomic and biochemical analyses that these changes affect the metabolic potential of the mouse gut microbiota. Furthermore, this trait is transmissible: colonization of germ-free mice with an 'obese microbiota' results in a significantly greater increase in total body fat than colonization with a 'lean microbiota'. These results identify the gut microbiota as an additional contributing factor to the pathophysiology of obesity. It has been suggested, therefore, that the obese microbiome has an increased capacity to harvest energy from the diet.

ELIGIBILITY:
Inclusion criteria

* 40 patients that refers to helicobacter pylori treatment
* Aged 20-60 years old
* 22 Kg/m2 ≤ BMI ≤ 30 Kg/m2
* Functional GI trace with permanent stool number
* Keeping on a permanent diet
* Written informed consent
* Stated availability throughout the study period
* Mental ability to understand and follow the protocol

Exclusion criteria

* Use of laxatives
* Confirmed GI tract infections or inflammatory bowel disease
* Any major chronic illness
* Pregnancy
* Participation in other clinical trials
* Use of oral or intravenous antibiotics during 8 weeks prior to recruitment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof., Study Director
Locations (1):
- The Unit of Clinical Nutrition, Tel Aviv, Israel